CLINICAL TRIAL: NCT06518863
Title: Elucidating the Relationship Between Ultra-Processed Food Consumption, Executive Function, and Hunger-Related Hormones
Brief Title: Ultra-Processed Foods and Executive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB-23-322-STW
Record Dates: First submitted 2024-05-16; First posted 2024-07-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-processed foods (Experimental): Participants are instructed to consume only ultra-processed foods for 3 days.
  Interventions: Behavioral: Education
- Unprocessed foods (Experimental): Participants are instructed to consume only unprocessed foods for 3 days.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Educational handouts on how to adhere to the corresponding diet.

SUMMARY:
The purpose of this study is to examine potential effects of a diet characterized by UPF on hunger-related hormones and executive function. It entails a two-arm, crossover, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55
* Willing to consume an entirely ultra-processed and entirely unprocessed diet for 3 days each (6 days in total)

Exclusion Criteria:

* Chronic disease that interferes with study-related activities
* Special diet that limits adherence to the intervention diets
* Visual impairment not corrected by glasses/contacts
* Pregnant or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Plasma ghrelin | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)

SECONDARY OUTCOMES:
Plasma active amylin | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Plasma C-peptide | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Plasma active glucagon-like peptide-1 (GLP-1) | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Plasma gastric inhibitory polypeptide (GIP) | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in pg/mL
Plasma glucagon | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Plasma insulin | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Plasma leptin | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Plasma monocyte chemoattractant protein-1 (MCP-1) | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Plasma pancreatic polypeptide (PP) | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Plasma peptide YY (PYY) | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Plasma secretin | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in picograms per milliliter (pg/mL)
Body mass | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in kilograms
Body mass index | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured in kilograms divided by meters squared
Percent fat mass | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured using a seca medical body composition analyzer (mBCA) 514 bioelectrical impedance scale, as a percentage
Body fat mass | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured using a seca medical body composition analyzer (mBCA) 514 bioelectrical impedance scale, in kilograms
Percent lean mass | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured using a seca medical body composition analyzer (mBCA) 514 bioelectrical impedance scale, as a percetange
Lean mass | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured using a seca medical body composition analyzer (mBCA) 514 bioelectrical impedance scale, in kilograms
Food addiction according to the Yale Food Addiction Scale Version 2.0 | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Presented as a symptom count (score range from 0-11, higher means more food addiction symptoms) and used to classify as "No," "Mild," "Moderate," or "Severe" food addiction
Behavioral Inhibition System/Behavioral Approach System Scale | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Score ranges from 20 to 80, with higher scores indicating greater behavioral inhibition and behavioral activation
Executive Function: Tower Test (Delis-Kaplan Executive Function System) | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Total Achievement Score (range=0-30, higher = higher executive function)
Executive Function: Color-Word Interference Test (Delis-Kaplan Executive Function System) | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Scaled inhibition/switching scores (score range=1-19, higher = higher executive function)
Ultra-processed food intake | Measured at three times: baseline, post-first diet arm (3 days), post-second diet arm (6 days)
  Measured as a percent of total calories, taken from 3-day diet records

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No